CLINICAL TRIAL: NCT00935441
Title: Effect of Nurse-Based, Protocol-Driven, Case-Management Utilizing Home Telemonitoring and Home HbA1c Measurement on Diabetes and Blood Pressure Outcomes
Brief Title: Effect of Case-Management Using Home Monitoring on Diabetes and Blood Pressure Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nacide Ercan-Fang, Principal Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4127-B
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; chronic care; case management; telemedicine
MeSH Terms: conditions — Diabetes Mellitus | interventions — Case Management

ARMS (2):
- Telemonitoring (Experimental): Case management with home telemonitoring for blood sugar and blood pressure plus home HbA1c measurement
  Interventions: Behavioral: case management with telemonitoring
- Usual case management (Active Comparator): Case management
  Interventions: Behavioral: usual case management

INTERVENTIONS:
Behavioral: case management with telemonitoring — telephone contact with a case manager, home telemonitoring equipment for blood sugar and blood pressure, home HbA1c measurement
  Arms: Telemonitoring
Behavioral: usual case management — telephone contact with a case manager
  Arms: Usual case management

SUMMARY:
This is a randomized trial designed to determine if adoption of the chronic care model in conjunction with nurse case management, home telemonitoring, and home HbA1c monitoring can improve glycemic control compared to patients receiving usual case management. We hypothesize that nurse case management, with home telemonitoring of blood sugars and home HbA1c measurement will result in additional improvements in glycemic control compared to isolated nurse case management. Specifically, the telemonitoring group will have an HbA1c 0.5% lower compared to usual nurse case management. Secondary aims include an additional 5 mmHg improvement in systolic blood pressure (among patients with hypertension at the time of enrollment), improved patient satisfaction with treatment, improved medication adherence, reduced incidence of hypoglycemia, and reduced case manager time in the telemonitoring/home HbA1c group compared with usual caes management. The study will enroll 460 diabetic patients with HbA1c values greater than 8.5%, age 75 years or younger, who have a active land-line for telephone communication. Patients will be enrolled and actively case managed for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at Minneapolis VAMC,
* Type 1 or 2 Diabetes,
* HbA1c >8.5%,
* active land-line telephone connection

Exclusion Criteria:

* Age >75 years,
* primary care provider unwilling to have patient enrolled,
* active dialysis,
* resident of assisted living facility,
* research participant in previous diabetes case management study,
* life expectancy <1 year,
* severe mental health condition,
* active substance abuse,
* pregnant or planning on becoming pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | 9 months after enrollment

SECONDARY OUTCOMES:
Systolic blood pressure control in patients with elevated blood pressure at baseline | 9 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VAMC, Minneapolis, Minnesota, United States